CLINICAL TRIAL: NCT06059274
Title: Evaluation of the Efficacy of an Anti-aging Repairing Serum Containing Hyaluronic Acid, Vitamin B5, Madecassoside and La Roche-Posay Thermal Spring Water
Brief Title: Anti-aging Repairing Serum: Efficacy and Tolerability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1718CBCL357-Serum
Record Dates: First submitted 2023-09-23; First posted 2023-09-28 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Anti-aging
Keywords: anti-aging; skin barrier; dermocosmetic; wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical serum (Experimental): An investigational topical serum containing hyaluronic acid, vitamin B5, madecassoside and La Roche-Posay Thermal Spring Water
  Interventions: Other: Topical serum

INTERVENTIONS:
Other: Topical serum — Participants are asked to apply the topical serum twice daily for 84 days.

SUMMARY:
The study aimed to evaluate the effectiveness and tolerability of a dermocosmetic serum containing hyaluronic acid, vitamin B5, madecassoside and La Roche-Posay Thermal Spring Water in reducing skin aging signs. The experimental clinical trial involved 34 participants aged 45 to 65 years who applied the serum twice a day for 84 days.

DETAILED DESCRIPTION:
This experimental, mono-centric, open clinical trial was conducted in accordance with the principles of Resolution 466/2012 of the Conselho Nacional de Saúde do Brasil, ethical principles from the Declaration of Helsinki (and subsequent modifications) and Good Clinical Practice (GCP).

Quality control was applied to each stage of data handling to ensure that clinical data were generated, collected, processed, analyzed and reported according to the protocol, Standard Operating Procedures (SOP) and requirement of GCP.

Descriptive Statistics: Quantitative parameters, or those that can be reasonably treated as such, were summarized using measures of central tendency as mean and median and dispersion measures as standard deviation at each time of evaluation. Quantitative variables were summarized using frequencies and percentages. For each parameter (clinical evaluation scores and parameters derived from the Primos®) and each region (frontal, periocular, peri-oral and neck), graphical representations of means ± 95% Confidence Interval (CI) were elaborated for visual assessment of evolution over time.

ELIGIBILITY:
Inclusion Criteria:

* phototype I to IV
* presenting wrinkles on the forehead and/or peri-orbital area with grade ≥ 2 and ≤4 according to "Skin Aging Atlas"
* participant has not used any anti-aging products or performed aesthetic procedures over the last three months

Exclusion Criteria:

* pregnant, breastfeeding or immune compromised woman
* participant with cutaneous marks or active dermatoses on the tested area that could interfere with the evaluation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Instrumental Assessment - Primos® Optical 3D | from baseline to Day 84
  The Primos® Optical 3D (Canfield) device in vivo allows the measurement and evaluation of wrinkles through the technique of fringed projection, based on digital mirrors (DMDTM: Digital Mirco mirror Devices) directly on the skin surface of the participants.
Clinical assessment through Visual Analog Scale (VAS) | from baseline to Day 84
  The dermatologist investigates the degree of roughness of the frontal, peri-orbital, peri-oral, neck and overall aspect according to the following parameters: number of wrinkles (no wrinkles / several wrinkles), wrinkles thickness (very thin wrinkle / very thick wrinkle), length of the wrinkle (very short wrinkle / very long wrinkle), depth of wrinkle (very superficial wrinkle / very deep wrinkle) on a line from 0 to 10.
Clinical assessment using the standard scale "Skin Aging Atlas" | from baseline to Day 84
  The dermatologist investigates the frontal, peri-orbital, peri-oral and neck regions, comparing the roughness observed in the research regions with the images presented in the Skin Aging Atlas, establishing, for each area, a degree of roughness, that made possible the evaluation in the different experimental times.

SECONDARY OUTCOMES:
Instrumental Assessment - VISIA-6® | from baseline to Day 84
  Standardized photographs with VISIA-6® are taken of the participants' right, left and front profiles using standard and cross-polarized lights.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, Principal Investigator — Centre International de Développement Pharmaceutique (CIDP)
Locations (1):
- CIDP Brasil, Rio de Janeiro, Brazil